CLINICAL TRIAL: NCT04391764
Title: Effect of Naltrexone in Achieving and Maintaining Abstinence From Alcohol in Patients With Cirrhosis- A Double Blind Randomized Controlled Trial.
Brief Title: Effect of Naltrexone in Achieving and Maintaining Abstinence From Alcohol in Patients With Cirrhosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-28
Record Dates: First submitted 2020-05-08; First posted 2020-05-18 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexone (Experimental): Naltrexone at a dose of 50 mg per day.
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Placebo tablets will be identical in size, colour, shape, and taste and will be given in a similar manner.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Naltrexone — Naltrexone at a dose of 50 mg per day
  Arms: Naltrexone
Drug: Placebo oral tablet — Placebo tablets will be identical in size, colour, shape, and taste and will be given in the similar manner.
  Arms: Placebo

SUMMARY:
The aim of the study is to study the safety and tolerability of Naltrexone in patients with Alcohol liver disease over a 12 week duration without liver related side effects. The project will be conducted at ILBS from March 2020 to February 2021. The concept is to estimate the usage of naltrexone and establish its safety in cirrhotics and study its effect on achieving and maintaining abstinence and in reducing lapses and relapses. Thereby reducing the progression of alcoholic liver disease as continued ethanol consumption is an important predictor in increasing overall morbidity and mortality.

All ALD patients will be included as per inclusion and exclusion criteria, after taking informed consent from the patient or their relatives. In case of any reactions, the drug will be stopped as per the study stopping rule.

After following the inclusion and exclusion criteria, ALD patients will be recruited into the study. It's a double blind RCT, hence both the patient and the investigator will be blinded and the drug will be issued by the trial co-ordinator after taking informed written consent and explaining the side effects. Naltrexone at a dose of 50 mg per day and placebo are included in the tablets. Placebo tablets will be identical in size, colour, shape, and taste. Naltrexone tablets will be entrusted to a family member to administer every dose and monitor for side effects.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive alcohol dependent cirrhotic aged between 18-60 yrs.
2. Fulfilling DSM - 5 criteria for alcohol use disorder (Association, 2013).

Exclusion Criteria:

1. Current Hepatic Encephalopathy
2. Total Bilirubin > 3 mg/dl.
3. Recent bleed.
4. Treatment with corticosteroids within the past 60 days.
5. Unwilling to participate.
6. Dependence on any other substance (except Nicotine).
7. Psychotic disorder requiring treatment/Suicidal tendency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving and maintaining alcohol abstinence at 12 weeks in both groups | 12 weeks

SECONDARY OUTCOMES:
Proportion of patients on Naltrexone without liver related adverse effects as compared to placebo | 12 weeks
Proportion of patients maintaining abstinence from alcohol at 6 months in both groups | 6 months
Proportion of patients maintaining abstinence from alcohol at 12 months in both groups | 12 months
difference in craving measures between groups at 4 weeks in both groups | 4 weeks
  OCDS (Obsessive-Compulsive Drinking Scale) scale will be use to measure the craving
difference in craving measures between both groups at 8 weeks. | 8 weeks
  OCDS (Obsessive-Compulsive Drinking Scale) scale will be use to measure the craving
difference in craving measures between both groups at 12 weeks. | 12 weeks
  OCDS (Obsessive-Compulsive Drinking Scale) scale will be use to measure the craving
difference in craving measures between both groups at 6 months. | 6 months
  OCDS (Obsessive-Compulsive Drinking Scale) scale will be use to measure the craving
difference in craving measures between both groups at 12 months. | 12 months
  OCDS (Obsessive-Compulsive Drinking Scale) scale will be use to measure the craving

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided